CLINICAL TRIAL: NCT00262587
Title: Elite Sport and Development of Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Imperial College London (Other); Anti Doping Danmark (Other); GlaxoSmithKline (Industry); The Research Foundation of Bispebjerg Hospital (Unknown); Ragnhild Ibsens Legat For Medicinsk Forskning (Other)
Responsible Party: Principal Investigator, Thomas Lund, MD, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-061; (KF) 01 262958
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Asthma
Keywords: Sport; Asthma; Treatment; Airway inflammation
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator): Placebo inhaler (sugar powder)
  Interventions: Drug: Placebo
- Seretide (Active Comparator): Seretide inhaler
  Interventions: Drug: Seretide

INTERVENTIONS:
Drug: Seretide — Combination of inhaled corticosteroids (250 microgr) and inhaled long-acting beta2-agonists (25 microgr)
  Arms: Seretide
Drug: Placebo — Inhaled sugar powder in a placebo inhaler
  Arms: Placebo

SUMMARY:
International studies have shown that elite athletes have a high prevalence of respiratory symptoms and asthma as compared to normal subjects. It is unclear whether the increased prevalence of asthma in elite athletes reflects "traditional asthma" or whether it is a special form of "sports asthma". The treatment of elite athletes with asthma seems to vary widely, and only a few studies have focused on the treatment of elite athletes with asthma. Further knowledge of the pathogenesis of sports asthma would lead to a greater understanding and better treatment of the condition. This study will investigate the type of airway inflammation in elite athletes and examine the effect of treatment with inhaled steroids in combination with long-acting beta-agonists versus placebo in the same group.

ELIGIBILITY:
Inclusion Criteria:

* Elite athletes
* Informed consent
* Doctor diagnosed asthma

Exclusion Criteria:

* Current smoker or more than 10 pack-years
* Pregnancy, breast feeding or planning pregnancy during the study.
* ICS within the last 4 weeks prior to visit 1.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2005-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Eucapnic voluntary hyperventilation (EVH) | End of study
Exhaled Nitric Oxide | End of study

SECONDARY OUTCOMES:
Respiratory symptoms | End of study
Lung function | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lund, MD, Principal Investigator — Respiratory and Allergy Research Unit, Department of Respiratory Medicine
Locations (1):
- Respiratory and Allergy Research Unit, Department of Respiratory Medicine, Bispebjerg Hospital, Copenhagen, Denmark